CLINICAL TRIAL: NCT06883786
Title: Interest of Virtual Reality Hypnosis to Decrease Anxiety, Pain, and Discomfort of Patients With Cancer Having to Undergo an Invasive Intervention
Brief Title: Effects of Virtual Reality Hypnosis on Anxiety, Pain and Comfort in Oncology Patients During a Port-catheter Placement Procedure
Acronym: VRH-PAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: HypnoVR (Industry); Centre Hospitalier Regional de Huy (Other); University hospital of Liège (Unknown)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD, Responsible of the Sensation and Perception Research Group, in the GIGA CONSCIOUSNESS department, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VRH-PAC
Record Dates: First submitted 2024-02-15; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality hypnosis (Experimental): The VRH session, called Aqua+© (120 Version 1.1, HypnoVR SAS, Strasbourg, France) It is an immersive and contemplative virtual experience combining music, sounds, and/or a vocal audio recording relating a hypnotic scenario and a 3D virtual video. The Aqua© VRH session follows the standard phases of hypnosis, beginning with induction, followed by suggestions, and ending with the exit of hypnosis.
  Interventions: Device: Virtual reality hypnosis
- Control (No Intervention): Usual care. Local anesthesia only.

INTERVENTIONS:
Device: Virtual reality hypnosis — Virtual reality hypnosis
  Arms: Virtual reality hypnosis

SUMMARY:
The port-catheter (PAC) is a longterm venous access device, frequently used in oncology patients. The PAC is an invasive technique, consisting of a reservoir surgically implanted in the chest wall or upper arm, and arm and a catheter. Patients can experience pain in the incision area after implantation, as well as anxiety before, during and after implantation. Virtual reality hypnosis (VRH) is an innovative technique delivering clinical hypnosis to patients through virtual reality (VR). The clinical applications of VRH are still little known. We will assess the anxiety, comofrt, pain perception and pain unpleasantness of 102 cancer patients scheduled to receive a PAC. The patients will be randomly divided into two groups. Thefirst group will benefit from the usual care for the placement of the PAC (i.e., local anaesthesia), while the second will benefit from the VRH in addition to the usual care. Pain perception, pain unpleasantness, anxiety, satisfaction, absorption, dissociation will be evaluated before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Low auditory and/or visual acuity precludes the use of the device.
* Head or face wounds precluding the use of the device.
* Schizophrenia, dissociative disorder or any other psychiatric disorder.
* Non-proficiency in French (Research language).
* Patient under 18 years old.
* Phobia of deep water.
* Dizziness.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Anxiety state | Before PAC intervention, immediately after PAC intervention
  Anxiety state will be assessed using a numerical rating scale (NRS) ranging from 0 (no anxiety) to 10 (worst anxiety ever).
Pain intensity | Before PAC intervention, immediately after PAC intervention
  Pain intensity will be assessed using a numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Pain unpleasantness | Before PAC intervention, immediately after PAC intervention
  Pain unpleasantness will be assessed using a numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Comfort | Before PAC intervention, immediately after PAC intervention
  Comfort will be assessed using a numerical rating scale (NRS) ranging from 0 (no comfort) to 10 (maximum comfort).

SECONDARY OUTCOMES:
Anxiety trait | From the day of the group assignment until beginning the PAC intervention, assessed up to two weeks
  The State-Trait Anxiety Inventory (STAI - Y) will be used to assess trait anxiety only. Originally this questionnaire has two parts one dedicated to assess state anxiety and another to assess the trait anxiety. Only the latter was used in this study. STAI - Y Trait contains 20 items with 4 response options (1 = almost never, 2 = sometimes, 3 = often, 4 = almost always). Total scores can range from 20 to 80, with higher scores indicating a higher level of anxiety.
Dissociation trait | From the day of the group assignment until beginning the PAC intervention, assessed up to two weeks
  The Dissociative Experience Scale is a self-reported questionnaire used to evaluate the presence, quantity, and type of dissociative experiences one might live in daily life. It consists of 28 items arranged on an analog scale (from 0 to 100% measuring the frequency of dissociative experiences), and the total score ranges from 0 to 100. There is a cutoff of 45 as a mean score to suggest a dissociative disorder. This questionnaire is not a diagnostic instrument; it is designed only for screening, but it can suggest that a specific clinical assessment is needed.
Dissociation state | From the day of the group assignment until completion of the PAC intervention, assessed up to two weeks
  Dissociation will be assessed using a numerical rating scale (NRS) ranging from 0 (no dissociation) to 10 (maximum dissociation).
Absorption trait | From the day of the group assignment until beginning the PAC intervention, assessed up to two weeks
  The Tellegen Absorption Scale consists of 34 true/false items , aiming to measure the absorption of a person, meaning the disposition for having episodes of a deep involvement that engage all the subject's resources (perceptual, imaginative, and cognitive). The total score range is from 0 to 34. The higher the score, the more one has a high propensity for absorption.
Absorption state | From the day of the group assignment until completion of the PAC intervention, assessed up to two weeks
  Absorption will be assessed using a numerical rating scale (NRS) ranging from 0 (no Absorption) to 10 (maximum Absorption).
Time perception | From the day of the group assignment until completion of the PAC intervention, assessed up to two weeks
  Time perception will be assessed with an open-ended question.
Immersion tendencies | From the day of the group assignment until beginning the PAC intervention, assessed up to two weeks
  Immersion propensity is the amount of sensory input the virtual reality system creates. Will be assessed with the Immersion Propensity questionnaire. The higher the score, the more one is immersed in the virtual environments.
Satisfaction of the participant | From the day of the group assignment until completion of the PAC intervention, assessed up to two weeks
  Satisfaction will be assessed using a numerical rating scale (NRS) ranging from 0 (dissatisfied) to 10 (best satisfaction ever).
Satisfaction of the surgeon | From the day of the group assignment until completion of the PAC intervention, assessed up to two weeks
  Satisfaction will be assessed using a numerical rating scale (NRS) ranging from 0 (dissatisfied) to 10 (best satisfaction ever).
Medication | During PAC intervention, 24 hours after PAC intervention, 48 hours after PAC, 7 days after PAC
  The medication will be collected in the medical record of the surgery.
Surgery duration | From the day of the group assignment until completion of the PAC intervention, assessed up to two weeks
  The duration of the surgery will be collected in the medical record of the surgery.
Fatigue | 24 hours after PAC intervention, 48 hours after PAC, 7 days after PAC
  Fatigue will be assessed using a numerical rating scale (NRS) ranging from 0 (no fatigue) to 10 (worst fatigue ever).

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - CHR de Huy, Huy, Liège
  - CHU of Liège, Liège, Liège